CLINICAL TRIAL: NCT00001496
Title: Establishment of Normal Breast Epithelial Cell Lines From Patients at High Risk for Breast Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960026; 96-C-0026
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-11

CONDITIONS: Breast Neoplasm; Hereditary Neoplastic Syndrome
Keywords: BRCA-1; Familial Breast Cancer; Breast Cell Culture; High Risk
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Syndromes, Hereditary; Breast Cancer, Familial

SUMMARY:
Women who are at high risk for breast cancer, either because of linkage to high risk breast and ovarian cancer families, or because of a carcinoma in the opposite breast, will be studied. Women will have a physical examination and mammography to ensure that no breast abnormalities are present. Eligible women will undergo biopsy of the breast to obtain normal breast tissue. Short-term cell cultures will be established from this tissue and early passages of the short-term cell lines will be stored. A bank of high risk normal mammary epithelial cells will be established. To further characterize the mammary epithelial cells in this population of women, cell cultures will subsequently be analyzed for their growth and metabolic properties, sensitivity to chemopreventive agents, steroid receptor characteristics, oncogene expression and regulation, and genetic changes.

DETAILED DESCRIPTION:
Women who are at high risk for breast cancer, either because of linkage to high risk breast and ovarian cancer families, or because of a carcinoma in the opposite breast, will be studied. Women will have a physical examination and mammography to ensure that no breast abnormalities are present. Eligible women will undergo biopsy of the breast to obtain normal breast tissue. Short-term cell cultures will be established from this tissue and early passages of the short-term cell lines will be stored. A bank of high risk normal mammary epithelial cells will be established. To further characterize the mammary epithelial cells in this population of women, cell cultures will subsequently be analyzed for their growth and metabolic properties, sensitivity to chemopreventive agents, steroid receptor characteristics, oncogene expression and regulation, and genetic changes.

ELIGIBILITY:
Women at high risk for breast cancer, either because they are a member of a high risk breast or ovarian cancer family, or because of a carcinoma of the opposite breast.

Normal mammogram within past 3 months.

No suspicious breast or axillary lesions on physical examination.

No major cardiopulmonary, hepatic or renal disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1996-01; Study Completion 2001-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Miki Y, Swensen J, Shattuck-Eidens D, Futreal PA, Harshman K, Tavtigian S, Liu Q, Cochran C, Bennett LM, Ding W, et al. A strong candidate for the breast and ovarian cancer susceptibility gene BRCA1. Science. 1994 Oct 7;266(5182):66-71. doi: 10.1126/science.7545954.
- [Background] Sgagias MK, Gagneton DC, Rosenberg SA, Danforth DN Jr. Cellular characterization and retroviral transduction of short-term breast cancer cells. J Immunother Emphasis Tumor Immunol. 1995 Feb;17(2):88-97. doi: 10.1097/00002371-199502000-00003. PMID 7647960
- [Background] Wooster R, Neuhausen SL, Mangion J, Quirk Y, Ford D, Collins N, Nguyen K, Seal S, Tran T, Averill D, et al. Localization of a breast cancer susceptibility gene, BRCA2, to chromosome 13q12-13. Science. 1994 Sep 30;265(5181):2088-90. doi: 10.1126/science.8091231.